CLINICAL TRIAL: NCT03118336
Title: Impact of Empaglifozine on Cardiac Ectopic Fat
Acronym: EMPACEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-39; 2016-003196-21 (EudraCT Number)
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator)
  Interventions: Drug: Empagliflozin 10Mg Tab
- empaglifozine group (Experimental)
  Interventions: Drug: Empagliflozin 10Mg Tab

INTERVENTIONS:
Drug: Empagliflozin 10Mg Tab — 1 tablet of 10 milligrams per bone 1 time a day during 12 weeks

SUMMARY:
There is substantial evidence supporting the fact that ectopic fat accumulation is an important contributor to type 2 diabetes complications and cardiovascular risk [1]. Epicardial adipose tissue (EAT), located between the myocardium and the visceral layer of the pericardium has been associated with atrial fibrillation and with coronary artery disease [2, 3] and its abundance predicts the number of cardiac events within 8 years [4]. In addition, myocardial steatosis has been shown to be an independent predictor of diastolic dysfunction [5] [6]. Furthermore, in type 2 diabetic patients, bariatric surgery can reduce cardiac ectopic fat accumulation and improve cardiac function [7] [8]. When added to standard care, 10 or 25 mg/d of empagliflozin, an inhibitor of sodium-glucose cotransporter 2 (iSGLT2), significantly reduces the risk of death, cardiovascular death, and hospitalisation for heart failure among individuals with type 2 diabetes and established cardiovascular disease when compared to placebo [9]. The mechanisms of empagliflozin-improved cardiovascular outcomes in type 2 diabetic patients at high risk of cardiovascular events are not known. We hypotheses that empaglifozin could modulate cardiac ectopic fat and cardiac metabolism in obese type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Type 2 diabetes based on the disease diagnostic criteria as described by the WHO,
* HbA1c > 7% and < 10 %
* Stable glucose-lowering therapy for at least 3 weeks before randomization
* Estimated glomerular filtration rate > 60/ml (MDRD)
* Signed informed consent form obtained prior to any study procedure

Exclusion Criteria:

* Evolutive or planned pregnancy during the six months
* Lactation
* Recent weight loss (>5% of body weight within one month),
* Treatment modifying adipose distribution such as corticoids
* Acute coronary syndrome or instable angina during the last 2 months,
* MRI contraindication (metal cardiac valve, pace maker, metal foreign body, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
cardiac morphology | 12 weeks
  magnetic resonance imaging
epicardial adipose tissue volume | 12weeks
  magnetic resonance imaging

SECONDARY OUTCOMES:
myocardial triglyceride | 12weeks
  proton magnetic resonance spectroscopy
hepatic triglyceride content | 12 weeks
  proton magnetic resonance spectroscopy
myocardial PCr/ATP ratio | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: anne dutour, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soghomonian A, Dutour A, Kachenoura N, Thuny F, Lasbleiz A, Ancel P, Cristofari R, Jouve E, Simeoni U, Kober F, Bernard M, Gaborit B. Is increased myocardial triglyceride content associated with early changes in left ventricular function? A 1H-MRS and MRI strain study. Front Endocrinol (Lausanne). 2023 Jun 22;14:1181452. doi: 10.3389/fendo.2023.1181452. eCollection 2023. PMID 37424866
- [Derived] Gaborit B, Ancel P, Abdullah AE, Maurice F, Abdesselam I, Calen A, Soghomonian A, Houssays M, Varlet I, Eisinger M, Lasbleiz A, Peiretti F, Bornet CE, Lefur Y, Pini L, Rapacchi S, Bernard M, Resseguier N, Darmon P, Kober F, Dutour A. Effect of empagliflozin on ectopic fat stores and myocardial energetics in type 2 diabetes: the EMPACEF study. Cardiovasc Diabetol. 2021 Mar 1;20(1):57. doi: 10.1186/s12933-021-01237-2. PMID 33648515